CLINICAL TRIAL: NCT04093882
Title: The Relevance of the Blood-brain Barrier to Cognitive Dysfunction and Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. med. Jochen Fiebach (Senior Physician) (Unknown)
Responsible Party: Principal Investigator, Oliver Peters, MD, Prof. dr. med. (Consultant Psychiatrist), Charite University, Berlin, Germany
Other Study IDs: BHSkog
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Blood Brain Barrier; Alzheimer Disease; Cognitive Dysfunction; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Cerebro-spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitive normal: Individuals who do not show clinical or neuropsychological deficits.
  Interventions: Diagnostic Test: Contrast agent enhanced MRI using Gadovist
- Mild cognitive impairment: Individuals who show deficits in neuropsychological test procedures but who do not exhibit substantial problems in daily life. Those individuals are part of the DELCODE cohort and were initially recruited in a memory clinic.
  Interventions: Diagnostic Test: Contrast agent enhanced MRI using Gadovist
- Dementia due to Alzheimer's disease: Individuals diagnosed with dementia due to Alzheimer's disease by relying on anamnesis, neuropsychological test results, results of MRI and biomarkers found in the cerebrospinal fluid. Those individuals are part of the DELCODE cohort and were initially recruited in a memory clinic.
  Interventions: Diagnostic Test: Contrast agent enhanced MRI using Gadovist

INTERVENTIONS:
Diagnostic Test: Contrast agent enhanced MRI using Gadovist — By using the contrast agent Gadovist we aim to visualize the blood-brain barrier. Furthermore, we aim to measure a newly developed biomarker of the blood-brain barrier in the cerebro-spinal fluid.

SUMMARY:
This study attempts to replicate the findings published in Nature Medicine by Nation and colleagues (2019). By using a large observational cohort (DZNE - Longitudinal Cognitive Impairment and Dementia Study; DELCODE) consisting of cognitively healthy individuals, individuals with subjective cognitive decline, mild cognitive impairment, and dementia due to Alzheimer's disease, an association between the blood-brain barrier and cognitive dysfunction is investigated. The integrity of the blood-brain barrier is investigated by using a novel MRI protocol as well as a novel biomarker in the cerebrospinal fluid.

ELIGIBILITY:
Inclusion criteria:

- ≥ 50 years with neuropsychologically confirmed no cognitive dysfunction, mild cognitive impairment or mild dementia

Exclusion cirteria:

* no current or prior history of any neurological or psychiatric condition, which might affect cognitive function
* no neurodegenerative disease other than AD
* specifically no extensive vascular white matter dementia or vascular dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A description of the study population is provided by DZNE - Longitudinal Cognitive Impairment and Dementia Study (DELCODE).
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Marker of blood-brain dysfunction using MRI | 1 day
  Dynamic T1 contrast enhanced sequence using Gadovist
Markers of blood-brain dysfunction using CSF | 1 day
  Platelet-derived growth factor receptor-β in CSF

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No